CLINICAL TRIAL: NCT00549640
Title: Efficacy of Methylphenidate for Treating Tobacco Dependence
Brief Title: Testing Methylphenidate for Smoking Abstinence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Richard D. Hurt, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-005407; 06-006284 (Other: Mayo Clinic IRB Number)
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Results first posted 2010-11-01 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Smoking
Keywords: nicotine dependence; tobacco dependence
MeSH Terms: conditions — Smoking; Tobacco Use Disorder | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylphenidate (Active Comparator): 54 mg Methylphenidate per day for 8 weeks. Allowing for a ramp up in the first two weeks (starting dose is 18 mg/day).
  Interventions: Drug: Methylphenidate
- Placebo (Placebo Comparator): non-active (sugar pill)designed to be a look-alike to the methylphenidate. Given at the same frequency and dosage look-alike to the active comparator (methylphenidate 54 mg)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — 54 mg Methylphenidate per day for 8 weeks. Allowing for a ramp up in the first two weeks (starting dose is 18 mg/day).
  Other Names: Methylphenidate, Osmotic Release methylphenidate (OROS-MPH)
  Arms: Methylphenidate
Drug: Placebo — non-active (sugar pill)designed to be a look-alike to the methylphenidate. Given at the same frequency and dosage look-alike to the active comparator (methylphenidate 54 mg)
  Arms: Placebo

SUMMARY:
Cigarette smoking continues to be a major public health problem. Tobacco dependence interventions, as recommended by the USPHS Clinical Practice Guideline are not effective for all smokers. A need exists for new medications to treat various aspects of tobacco dependence, such as the reinforcing effects of nicotine, relief of nicotine withdrawal symptoms and prevention of early relapse. The neurobiology of the effect of methylphenidate is similar to that of the reinforcing effects of nicotine. In a small previous study, methylphenidate was reported to improve nicotine withdrawal symptoms and short term quit rates. Methylphenidate is well tolerated, has low abuse potential, and is less expensive compared to other tobacco dependence interventions. ConcertaTM, a long acting preparation of methylphenidate, is administered once a day, has similar bioavailability as the generic drug administered 3 times a day and has an overall similar or improved efficacy compared to generic methylphenidate. We plan to obtain preliminary efficacy data in a randomized, placebo-controlled phase II study assessing the effect of methylphenidate in cigarette smokers for increasing 7-day point prevalence smoking abstinence at end of treatment and 7-day point prevalence and prolonged smoking abstinence at 6-months. Critical and systematic evaluations of newer, innovative, and well-tolerated treatments to help treat tobacco use and dependence will provide a wider choice of therapeutic agents to smokers wishing to become abstinent from tobacco use.

DETAILED DESCRIPTION:
Once enrolled in study, the subject will be put in one of 2 groups by chance (as in the flip of a coin). They will either receive methylphenidate or a placebo. Everyone in study will receive nicotine dependence counseling based on the intervention manual "Smoke Free and Living It". Everyone will be asked to complete weekly study visits for 8 weeks and one follow-up phone call at week 16 and a final study visit at week 24. The target quit day is the day after visit 4 (week 2 + 1 day). In the first two weeks after starting study medication they will slowly build up to 3 pills a day. For weeks 2 through 8 they will continue to take 3 pills a day.

ELIGIBILITY:
Inclusion Criteria:

1. Are between 18 to 65 years of age
2. Have smoked cigarettes daily for the past 6-months and are currently smoking > 10 cigarettes/day
3. Are willing to make an attempt to stop smoking
4. Are able to participate fully in all aspects of the study
5. Have been provided with, understand, and have signed the informed consent

Exclusion Criteria:

1. Have clinically significant levels of current depression as assessed by CESD and determined by the physician; or have a life-time diagnosis of bipolar disorder, schizophrenia or dementia as determined by physician investigator
2. Are currently (in previous 30 days) using any tobacco treatment program (i.e., behavioral therapy, nicotine replacement therapy, bupropion SR, varenicline, clonidine or nortriptyline)
3. Have used an investigational drug within the 30 days prior to enrolling in this study
4. Alcohol or drug abuse or dependence within the past year as assessed by the study investigators using CAGE questionnaire and the Drug Abuse Screening Test 20 (DAST-20)
5. Are pregnant, lactating, or of child bearing potential, likely to become pregnant during the medication phase and not willing to use contraception. The following birth control measures are acceptable: approved hormonal contraceptive medications or devices, approved intra-uterine contraceptive devices, the use of two combined barrier methods (diaphragm with spermicide or condom with spermicide), birth control pills, injections, intrauterine device [IUD], abstinence, or surgical sterilization of subject or of monogamous partner.
6. Have a history of any major cardiovascular event in the past 6-months including unstable angina, acute MI or coronary angioplasty
7. Have clinically significant acute or chronic, progressive or unstable neurologic (dementia, delirium or seizure disorder), hepatic, renal, cardiovascular, respiratory or metabolic disease that would limit participation in the study
8. Are currently on the following prescribed medications known to interact with methylphenidate and not able to stop the medication during the study period: stimulants, warfarin, anticonvulsants, antidepressants, antipsychotics, monoamine oxidase inhibitors, clonidine, theophylline and pseudo-ephedrine
9. Uncontrolled hypertension (>160/100) or tachycardia (Heart rate >110)
10. Have another house-hold member or relative participating in the study
11. Have known allergy to methylphenidate or its constituents
12. Have a specific medical condition where use of methylphenidate is contraindicated: narrow angle glaucoma, motor tics, family history or diagnosis of Tourette's syndrome, and history of GI obstruction (including history of strictures, adhesions, or abdominal surgery)
13. have an ECG with significant arrhythmias or abnormal conduction, which in the opinion of the physician investigator preclude participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D. Hurt, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Hurt RD, Ebbert JO, Croghan IT, Schroeder DR, Sood A, Hays JT. Methylphenidate for treating tobacco dependence in non-attention deficit hyperactivity disorder smokers: a pilot randomized placebo-controlled trial. J Negat Results Biomed. 2011 Jan 28;10:1. doi: 10.1186/1477-5751-10-1. PMID 21276244

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study began on 03/10/08 and the final subject was randomized to study drug on 11/4/08. All subjects were recruited at Mayo Clinic in Rochester, MN.
Pre-assignment Details: After obtaining consent, subjects were screened for study inclusion. If they passed study entry criteria, they were randomized to study. All randomized subjects were included in the analysis.
Groups:
- Methylphenidate: osmotic-release methylphenidate (OROS-MPH) at a dose of one 18 mg tablet a day with a dose escalation schedule in the first 2 weeks to achieve a maximum dose of 54 mg (three 18 mg tablets once daily)
- Placebo: Look alike placebo pill with same dosing schedule as active methylphenidate
Period: Overall Study
Arm/Group | Methylphenidate | Placebo
Started | 40 | 40
Completed | 22 (For the primary endpoint, subjects who discontinued participation were assumed to be smoking.) | 24
Not Completed | 18 | 16
Not completed — Withdrawal by Subject | 6 | 12
Not completed — Adverse Event | 5 | 0
Not completed — Lost to Follow-up | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylphenidate | Placebo | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 39 | 79
  >=65 years | 0 | 1 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 35.6 (11.0) | 38.0 (11.9) | 36.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 26 | 46
  Male | 20 | 14 | 34
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80
Cigarettes Per Day [Mean (Standard Deviation); unit: cigarettes per day] — Self-reported number of cigarettes smoked per day
  cigarettes per day | 19.7 (7.4) | 20.8 (8.2) | 20.2 (7.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Biochemically Confirmed to be Abstinent From Smoking at End of Treatment.
Description: Number of subject who self report no smoking in the last 7 days (7-day point prevalence)at the end of the medication phase (week 8) and are biochemically confirmed (expired carbon monoxide <= 8 ppm)
Time Frame: 8 weeks
Population: Intention to Treat. subjects with missing information were assumed to be using tobacco.
Measure: Number; unit: participants
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 40 | 40
participants | 1 | 4
Statistical Analysis 1: Comparison: Methylphenidate vs Placebo; Test type: Superiority or Other; p = 0.973, Fisher Exact; 1-tailed

2. Primary Outcome: Number of Subjects Biochemically Confirmed to be Abstinent From Smoking at End of Study
Description: Number of subject who self report no smoking in the last 7 days (7-day point prevalence)at the end of study (week 24) and are biochemically confirmed (expired carbon monoxide <= 8 ppm)
Time Frame: 6 months
Population: Intention to treat (ITT). subject who discontinued study participation were counted as using tobacco.
Measure: Number; unit: participants
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 40 | 40
participants | 4 | 3
Statistical Analysis 1: Comparison: Methylphenidate vs Placebo; Test type: Superiority or Other; p = 0.500, Fisher Exact; 1 tailed test

3. Secondary Outcome: The Change in the Average Nicotine Withdrawal Symptom Score From Baseline to 14 Days Post Target Quit Date.
Description: The average composite nicotine withdrawal score (using Minnesota Nicotine Withdrawal Scale) change from baseline for the first 14 days following target quit date. Scale scores range from 0 (none) to 4 (severe).
Time Frame: baseline and 14 days
Population: Analysis was restricted to subjects who had diary information available for the first 14 days following target quit date
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 27 | 37
units on a scale | 0.28 (0.42) | 0.24 (0.35)
Statistical Analysis 1: Comparison: Methylphenidate vs Placebo; Test type: Superiority or Other; p = 0.65, t-test, 2 sided; For each subject, the average daily withdrawal score for the 14 days following target quit date was calculated and expressed as a change from baseline
Statistical Analysis 2: Comparison: Methylphenidate vs Placebo; Test type: Superiority or Other; p = 0.79, Mixed Models Analysis; analysis performed using daily scores

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for 8 weeks of study medication. Serious adverse events were collected for the duration for the duration of the study period (6 months)
Arm/Group | Methylphenidate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 1/40
Other Adverse Events (participants affected / at risk) | 17/40 | 5/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methylphenidate (N=40) | Placebo (N=40)
hospitalization (General disorders) | 0 | 1 — hospitalization following overdose of alcohol and prescription drugs.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methylphenidate (N=40) | Placebo (N=40)
Restless (Nervous system disorders) | 5 | 2
Insomnia (General disorders) | 5 | 0
Headache (Nervous system disorders) | 3 | 1
Anorexia (Psychiatric disorders) | 3 | 0
vivid dreams (General disorders) | 2 | 1
nausea (Gastrointestinal disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No